CLINICAL TRIAL: NCT01605422
Title: Effect of Dietary Pulses on Acute Postprandial Glycemia and Food Intake Regulation: A Systematic Review and Meta-analyses
Brief Title: Meta-analyses of the Effect of Dietary Pulses on Acute Postprandial Metabolic Control
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: John Sievenpiper (Other)
Collaborators: Pulse Canada (Other); Canada Research Chairs Endowment of the Federal Government of Canada (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, John Sievenpiper, Adjunct Research Fellow, University of Toronto
Organization: University of Toronto (Other)
Other Study IDs: PC 2011 KRS
Record Dates: First submitted 2012-05-18; First posted 2012-05-24 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes; Prediabetes; Dysglycemia; Overweight; Obesity; Metabolic Syndrome; Cardiovascular Disease
Keywords: Systematic review and meta-analysis; Evidence-based medicine (EBM); Evidence-based nutrition (EBN); Clinical practice guidelines; Clinical trials; Dietary pulses; legumes; Beans, peas, chickpeas, lentils; glycemic index; postprandial glycemia; insulin resistance; body weight; appetite; food intake regulation; satiety; satiation
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Overweight; Obesity; Metabolic Syndrome; Cardiovascular Diseases; Insulin Resistance; Body Weight

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Dietary pulses — beans, peas, chickpeas, lentils in whole or flour form

SUMMARY:
Dietary pulses (beans, peas, chickpeas, and lentils), more commonly known as "legumes", are generally recognized as healthy components of the diet. Canada's Food Guide encourages consumptions of meat alternatives, such as beans "more often"; and the dietary guidelines for Americans both recommend consumption of 3 cups of legumes per week. However, there remains insufficient information on the usefulness of these foods in protecting heart health. To improve evidence-based guidance for dietary pulse recommendations, the investigators propose to conduct a systematic review of the effect of dietary pulse consumption on after-meal blood sugar levels, appetite, and food intake regulation to help explain their mechanism for improving longterm blood sugar and body weight control. The systematic review process allows the combining of the results from many small studies in order to arrive at a pooled estimate, similar to a weighted average, of the true effect. The investigators will be able to explore whether eating pulses has different effects between men and women, in different age groups and background disease states, and whether or not the effect of pulses depends on the dose and background diet. The findings of this proposed knowledge synthesis will help improve the health of Canadians through informing recommendations for the general public, as well as those at risk of heart disease and diabetes.

DETAILED DESCRIPTION:
Background: Pulses, including dry peas, beans, lentils and chickpeas, are a rich source of a number of healthy dietary components including dietary fiber, low glycemic index carbohydrate, vegetable protein and polyphenolics. To support health claims and evidence-based dietary guidelines, it is important to establish whether the glycemic control and weight loss benefits observed with dietary pulses are attributable to their proposed mechanism-of-action, whereby they reduce acute postprandial excursions in glycemia and contribute to satiety and decreased intake at subsequent meals.

Objectives: The objective of this project is to conduct two systematic reviews and meta-analyses of the effect of dietary pulse consumption on acute postprandial metabolic endpoints: (1) postprandial glycemia and (2) food intake regulation.

Design: The planning and conduct of the proposed meta-analyses will follow the Cochrane handbook for systematic reviews of interventions. The reporting will follow the Preferred Reporting Items for Systematic reviews and Meta-Analyses (PRISMA) guidelines.

Data sources: MEDLINE, EMBASE, CINAHL and The Cochrane Central Register of Controlled Trials will be searched using appropriate search terms.

Study selection: Acute, single bolus controlled feeding trials that investigate the effect of isocaloric exchange of dietary pulses for other carbohydrate foods on cardiometabolic risk outcomes in humans will be included. Studies that have a chronic feeding design, lack a control, or report comparisons not matched for available carbohydrate will be excluded.

Data extraction: Independent investigators (≥2) will extract information about study design, sample size, subject characteristics, pulse form, dose, follow-up, and the composition of the background diets. Mean±SEM values will be extracted for all outcomes. Standard computations and imputations will be used to derive missing variance data. Risk of bias and study quality will be assessed using the Cochrane Risk of Bias Tool and the Heyland Methodological Quality Score (MQS), respectively.

Outcomes: Each analysis will assess a different set of endpoints related to acute postprandial metabolic control: (1) postprandial glycemia (area under the curve [AUC], GI) and (2) food intake regulation (subjective appetite scores, 2nd meal intake).

Data synthesis: Separate pooled analyses will be conducted for each area of metabolic control using the Generic Inverse Variance method with random effects models. Random-effects models will be used even in the absence of statistically significant between-study heterogeneity, as they yield more conservative summary effect estimates in the presence of residual heterogeneity. Paired analyses will be applied to all crossover trials. Heterogeneity will be tested by Cochrane's Q and quantified by I2. Sources of heterogeneity will be explored by sensitivity and subgroup analyses. A priori subgroup analyses will include disease status, duration of test, pulse type, pulse dose, study design, study quality, baseline values, and change in fat, protein, and dietary fibre intake. Standard GI methodology compliance will be another a priori sungroup analysis for the postprandial glycemia analyses only. Significant unexplained heterogeneity will be investigated by additional post hoc subgroup analyses (e.g. age, sex, level of feeding control [metabolic, supplemented, dietary advice], washout in crossover trials, energy balance of the background diet, composition of the background diet [total % energy from fat, carbohydrate, protein], change in cholesterol intake, change in glycemic index, etc.). Meta-regression analyses will assess the significance of subgroups analyses. Publication bias will be investigated by the inspection of funnel plots and application of Egger's and Begg's tests.

Knowledge translation plan: Results will be disseminated through traditional means such as interactive presentations at local, national, and international scientific meetings and publication in high impact factor journals. Innovative means such as webcasts with e-mail feedback mechanisms will also be used. Knowledge Users will act as knowledge brokers networking among opinion leaders and different adopter groups to increase awareness at each stage. Four Knowledge Users will also participate directly as members of nutrition guidelines committees. Target adopters will include the clinical practice, public health, industry, research communities, and patient groups. Feedback will be incorporated and used to guide analyses and improve key messages at each stage.

Preliminary findings: We conducted a systematic review and meta-analysis of the effect of dietary pulses on glycemic control in 41 controlled feeding trials. We found that pulses alone or in low-glycemic index or high-fibre diets improved markers of glycemic control. Although the improvement was clinically significant, it came at the expense of substantial inter-study heterogeneity. Knowledge translation from this preliminary project has already begun. It has provided a rationale for a large trial of the effect of pulses in type 2 diabetes to address some of the identified sources of heterogeneity and is being used in the development of the 2013 CDA Clinical Practice Guidelines (CPG) for Nutrition Therapy.

Significance: The proposed project will demonstrate that the improvement in longterm glycemic control seen in our previous systematic review and meta-analysis of longterm randomized controlled feeding trials of pulses can be attributed to acute reductions in postprandial glycemia, reductions in appetite, and decreased intake at subsequent meals. This demonstration will aid in knowledge translation related to the effects of dietary pulses on cardiometabolic risk, strengthening the evidence-base for dietary recommendations and health claims and improving health outcomes through informing healthcare providers and patients, stimulating industry innovation, and guiding future research.

ELIGIBILITY:
Inclusion Criteria:

* dietary trials in humans
* acute, single bolus feeding
* control matched for available carbohydrate
* viable endpoint data

Exclusion Criteria:

* non-human studies
* chronic feeding
* lack of a suitable control (not matched for available carbohydrate)
* no viable endpoint data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Varied
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-09 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Effect of pulse consumption on post-prandial glycemia in acute, single bolus controlled feeding trials. | Up to 1.5-years
  Area under the curve [AUC], glycemic index (GI)
Effect of pulse consumption on satiety in acute, single bolus controlled feeding trials. | Up to 1.5-years
  Subjective appetite scores, 2nd meal intake

CONTACTS AND LOCATIONS:
Overall Officials: John L Sievenpiper, MD, PhD, Study Director — Department of Pathology and Molecular Medicine, McMaster University and Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital; Russell J de Souza, ScD, RD, Study Director — Department of Epidemiology and Biostatistics, McMaster University and Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital; David JA Jenkins, MD, PhD, DSc, Principal Investigator — Department of Nutritional Sciences and Medicine, University of Toronto and Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital; Cyril WC Kendall, PhD, Study Director — Department of Nutritional Sciences, University of Toronto and College of Pharamcy and Nutrition, University of Saskatchewan
Locations (1):
- The Toronto 3D (Diet, Digestive tract and Disease) Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Micheal's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Sievenpiper JL, Kendall CW, Esfahani A, Wong JM, Carleton AJ, Jiang HY, Bazinet RP, Vidgen E, Jenkins DJ. Effect of non-oil-seed pulses on glycaemic control: a systematic review and meta-analysis of randomised controlled experimental trials in people with and without diabetes. Diabetologia. 2009 Aug;52(8):1479-95. doi: 10.1007/s00125-009-1395-7. Epub 2009 Jun 13. PMID 19526214
- [Result] Li SS, Kendall CW, de Souza RJ, Jayalath VH, Cozma AI, Ha V, Mirrahimi A, Chiavaroli L, Augustin LS, Blanco Mejia S, Leiter LA, Beyene J, Jenkins DJ, Sievenpiper JL. Dietary pulses, satiety and food intake: a systematic review and meta-analysis of acute feeding trials. Obesity (Silver Spring). 2014 Aug;22(8):1773-80. doi: 10.1002/oby.20782. Epub 2014 May 13. PMID 24820437